CLINICAL TRIAL: NCT06494566
Title: Diet Supplementation of Omega-3 Fatty Acids After Surgical Treatment of Obesity: a Randomized Clinical Trial
Brief Title: Omega-3 Supplementation After Surgical Treatment of Obesity
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 10311419.5.0000.5333
Record Dates: First submitted 2019-07-22; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Obesity
Keywords: Sarcopenia; Lipid profile; Bariatric surgery; Metabolic surgery
MeSH Terms: conditions — Obesity; Sarcopenia | interventions — Docosahexaenoic Acids; Mineral Oil

STUDY DESIGN:
Intervention Model Description: Randomized, Double-blind, Placebo-controlled, Multicenter, CONSORT oriented study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized in blocks of two participants, at a 1:1 ratio, for the two groups of treatment. For every two participants, there will be one block. The number of each block will be hold in a nontransparent, seriated, sealed envelope. Intervention capsules will be opaque and stored in identical containers by a single investigator, who will not take part in data collection or analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Omega-3 (Active Comparator): Omega-3 2000mg (940mg of EPA and 660mg of DHA) in gastro resistant capsule by mouth once a day for 90 days, starting on day sixteen after surgery.
  Interventions: Dietary Supplement: Omega-3
- Placebo (Placebo Comparator): Mineral oil capsule by mouth once a day for 90 days, starting on day sixteen after surgery.
  Interventions: Dietary Supplement: Mineral Oil

INTERVENTIONS:
Dietary Supplement: Omega-3 — Omega-3 capsule
  Arms: Omega-3
Dietary Supplement: Mineral Oil — Mineral Oil Capsule
  Arms: Placebo

SUMMARY:
The study evaluates diet supplementation of Omega-3 fatty acids after surgical treatment of obesity in adults. Half participants will receive diet supplementation of Omega-3 fatty acids, while the other half will receive placebo.

DETAILED DESCRIPTION:
Omega-3 fatty acids has been related to immunomodulation and antioxidant action. Diet supplementation of Omega-3 fatty acids after surgical treatment of obesity may help stabilize protein catabolism, reduce peroxidative damage, and improve lipid profile.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30kg/m2
* Candidate to bariatric and metabolic surgery

Exclusion Criteria:

* Use of Omega-3
* Contraindication to bioimpedance analysis
* Uso of steroids, non steroidal inflammatory drugs, immunomodulators or antibiotics
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Weight | Assessment points: first and last preoperative nutritional assessment, fifteen days and three and a half months after surgery.
  Measurement with digital scale, patient standing, barefoot. kilograms (kg)
Height | Points of evaluation: first and last preoperative nutritional assessment, fifteen days and three and a half months after surgery.
  Height measurement, patient standing, barefoot. Unit of measurement: meters (m).

SECONDARY OUTCOMES:
Manual Grip Strength | Assessment points: first and last preoperative nutritional assessment, fifteen days and three and a half months after surgery.
  Best of three handgrip strength measurements, patient seated, arm supported. Unit of measurement: kilograms-force (kgf).
6-Minute Walk Test | Points of evaluation: first and last preoperative nutritional assessment, fifteen days and three months and medium after surgery.
  Walking with measurements of distance covered. Units of measurement: meters.
Electrical Bioimpedance - Percentage of muscle mass | Assessment points: first and last preoperative nutritional assessment, fifteen days and three and a half months after surgery.
  Electrical bioimpedance scale measurement. Unit of measurement: percentage (%).
Electrical Bioimpedance - Body fat percentage | Assessment points: first and last preoperative nutritional assessment, fifteen days and three and a half months after surgery.
  Electrical bioimpedance scale measurement. Unit of measurement: percentage (%).

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Irmandade Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Instituto de Cardiologia, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No